CLINICAL TRIAL: NCT03122938
Title: Effect of Daily Bovine Lactoferrin Supplementation on Fetal Development and Iron Metabolism in Healthy Pregnant Women: A Randomized Double-blind Controlled Trial
Brief Title: Lactoferrin Supplementation and Iron Metabolism in Healthy Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beingmate Baby & Child Food Co Ltd . (Other)
Collaborators: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RD02914009A
Record Dates: First submitted 2016-08-20; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Iron-deficiency Anemia
Keywords: lactoferrin; Iron Metabolism; iron-deficiency anemia; pregnant women; fetal development
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Food, Formulated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactoferrin Group (Experimental): lactoferrin-supplemented formula
  Interventions: Dietary Supplement: lactoferrin-supplemented formula
- Control Group (Placebo Comparator): formula without lactoferrin supplementation
  Interventions: Dietary Supplement: formula without lactoferrin supplementation

INTERVENTIONS:
Dietary Supplement: lactoferrin-supplemented formula — Subjects consume lactoferrin-supplemented formula (85mg lactoferrin per 100g) 3 times a day (81g totally).
  Other Names: Beingmate Nursing Mommy Formula
  Arms: Lactoferrin Group
Dietary Supplement: formula without lactoferrin supplementation — Subjects consume formula without lactoferrin supplementation (<6mg lactoferrin per 100g formula) 3 times a day (81g totally).
  Other Names: Beingmate Nursing Mommy Formula
  Arms: Control Group

SUMMARY:
To assess the effects of a lactoferrin supplemented formula on fetal development , iron metabolism and immunity in healthy pregnant women. One hundred and twenty healthy pregnant women (24<gestational weeks<26) are enrolled and randomly assigned to lactoferrin-supplemented formula group (active group) or normal formula group (control group, without lactoferrin supplementation). Subjects allocated in active group consume lactoferrin supplemented formula (85mg lactoferrin per 100g) 3 times a day (81g totally), while those in control group consume formula without lactoferrin supplementation (<6mg lactoferrin per 100g formula) according to the same schedule. Routine blood test including hemoglobin and serum ferritin, and food frequency questionnaire-based review and 24h*3 dietary record are performed every 4 weeks during intervention until delivery. Body weight of newborns are recorded after delivery. The differences in iron deficiency anemia morbility of pregnant women and anthropometric measurements of newborns between groups would be analyzed after completion of this study.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women with gestational weeks between 24 and 26;
* with hemoglobin concentration > 110g / L;
* without indication of abortion;
* without infectious disease or hereditary disease;
* without iron supplementation before enrollment.

Exclusion Criteria:

* with red blood count <3.5*10^12/L，hemoglobin concentration<110g/L or serum ferritin <20 μg/L；
* diagnosed with gestational diabetes mellitus;
* enrolled in other intervention study within past 1 month.

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
iron-deficiency anemia morbility of pregnant women | every 4 weeks during intervention, namely 28th gestational weeks, 32nd gestational weeks, 36th gestational weeks and the day of delivery.

SECONDARY OUTCOMES:
iron metabolism of pregnant women | every 4 weeks during intervention, namely 28th gestational weeks, 32nd gestational weeks, 36th gestational weeks and the day of delivery.
  hemoglobin concentration and serum ferritin concentration
fetal growth | the day of delivery, recorded by nurse.
  body weight of newborns
fetal growth and development | the day of delivery,recorded by nurse immediately
  body length of newborns
fetal development | the day of delivery, measured and recorded by nurse.
  head circumference

CONTACTS AND LOCATIONS:
Overall Officials: Fengbing Liang, Ph.D, Principal Investigator — Zhejiang University
Locations (1):
- Sir Run Run Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Available when oversight authorities require.